CLINICAL TRIAL: NCT03004313
Title: Structural and Molecular Neuroplasticity in Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Alexandre DaSilva, DDS, MS, Principal Investigator, Director of Headache and Orofacial Pain Effort, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00027383
Record Dates: First submitted 2011-08-30; First posted 2016-12-28 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Migraine
Keywords: migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Migraine (Experimental): 20 subjects experiencing 1-14 migraines per month will undergo the following:
  * Blood and urine samples will be collected
  * Complete a series of questionnaires; some of which will be completed daily
  * Quantitative Sensory Test (QST)will be performed
  * Magnetic Resonance Imaging (MRI)
  * PET imaging (during and outside of a migraine attack)
  Interventions: Procedure: Pet Scan; Procedure: MRI scan; Procedure: Quantitative Sensory Testing (QST)
- Healthy (Active Comparator): 20 healthy subjects will undergo the following:
  * Blood and urine samples will be collected
  * Complete a series of questionnaires; some of which will be completed daily
  * Quantitative Sensory Test (QST)will be performed
  * Magnetic Resonance Imaging (MRI)
  * PET imaging
  Interventions: Procedure: Pet Scan; Procedure: MRI scan; Procedure: Quantitative Sensory Testing (QST)

INTERVENTIONS:
Procedure: Pet Scan — Subjects will undergo Pet Scanning for 90 minutes
Procedure: MRI scan
Procedure: Quantitative Sensory Testing (QST)

SUMMARY:
The main purpose of this study is to integrate novel MRI techniques with positron emission tomography(PET) for the study of structural and molecular neuroplasticity in the brain of migraineurs, and its clinical association with changes in pain perception and modulation (e.g. allodynia). We will attempt to acquire images of the brain that may, in the future, assist doctors in better understanding how pain is felt and regulated in migraine sufferers.

DETAILED DESCRIPTION:
To investigate interictal opioid receptor (MOR) binding potential (BPND) changes in migraineurs as compared to age/gender-matched healthy controls. To demonstrate that frequency of the headache attacks and severity of cutaneous allodynia levels in migraineurs experienced over multiple attacks are correlated with levels of MOR BPND in specific brain regions. To investigate whether dysfunction of the pain regulatory endogenous opioid system of migraineurs is correlated with changes in the gray matter thickness in cortical areas associated with pain perception and modulation.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-45 years of age
* Between 1-14 migraine attacks per month or healthy

Exclusion Criteria:

* Cannot be taking daily migraine medication
* Healthy subjects cannot be taking hormonal birth control pills or other medication
* Cannot have chronic pain or a neurologic/psychiatric disorder such as: multiple sclerosis and bipolar disorder.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Level of mu-opioid receptor binding potential in the brain of episodic migraineurs during and outside the headache attack and compared to healthy controls. | 90 min PET scan

SECONDARY OUTCOMES:
Correlation of migraine attack severity in migraineurs with mu-opioid receptor binding potential | 90 min PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre DaSilva, DDS, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan - Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Jassar H, Nascimento TD, Kaciroti N, DosSantos MF, Danciu T, Koeppe RA, Smith YR, Bigal ME, Porreca F, Casey KL, Zubieta JK, DaSilva AF. Impact of chronic migraine attacks and their severity on the endogenous mu-opioid neurotransmission in the limbic system. Neuroimage Clin. 2019;23:101905. doi: 10.1016/j.nicl.2019.101905. Epub 2019 Jun 18. PMID 31279240